CLINICAL TRIAL: NCT02780674
Title: A Phase 1, Randomized, Blinded, Single-Dose, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of MEDI7734 in Type I Interferon-Mediated Autoimmune Diseases
Brief Title: A Phase 1 Study of MEDI7734 in Type I Interferon-Mediated Autoimmune Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6080C00001
Record Dates: First submitted 2016-05-03; First posted 2016-05-23 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Dermatomyositis, Polymyositis, Sjogren's, SLE, SSc
Keywords: Polymyositis, dermatomyositis, Sjogren's syndrome, SLE, SSc
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Sjogren's Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI7734 (Active Comparator): Three subjects (cohort 1) and six subjects (cohort 2-5) will receive MEDI7734 for a total of 27 subjects.
  Interventions: Biological: MEDI7734
- Placebo (Placebo Comparator): One subject (cohort 1) and two subjects (cohort 2-5) will receive placebo, for a total of 9 subjects.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI7734 — Three subjects (cohort 1) and six subjects (cohort 2-5) will receive MEDI7734 for a total of 27 subjects.
  Arms: MEDI7734
Biological: Placebo — One subject (cohort 1) and two subjects (cohort 2-5) will receive placebo, for a total of 9 subjects.
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of escalating, single subcutaneous doses of MEDI7734 in adult subjects with type I interferon-mediated autoimmune diseases.

DETAILED DESCRIPTION:
MEDI7734 is a human monoclonal antibody that binds to and causes temporary depletion of plasmacytoid dendritic cells (pDCs), a type of white blood cell. The objectives of this study are to evaluate the safety, drug levels, and pDC levels in subjects who are given a single injection of MEDI7734 or a placebo.

The study will be conducted in subjects with at least one of the five following autoimmune diseases: dermatomyositis, polymyositis, Sjogren's syndrome, systemic lupus erythematosus, or systemic sclerosis.

After a screening period, subjects will be randomized in a 3:1 ratio to receive a single dose of MEDI7734 or matching placebo, administered as a subcutaneous (under the skin) injection. After that, subjects will be evaluated periodically at the study site over at least the next 85 days.

Study acquired from Horizon in 2024. Originally Viela Bio was the sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18-65 years old
2. Diagnoses of dematomyositis, polymyositis, Sjogren's syndrome, systemic lupus erythematosus and/or systemic sclerosis based on standard criteria.
3. Weight 40-120kg
4. Stable disease such that in the opinion of the investigator it is unlikely that a change in subject's therapeutic regimen would be required during the subsequent 3 months.

Key Exclusion Criteria:

1. History of a hypersensitivity reaction or anaphylaxis to a previous mAb or human immunoglobulin therapy.
2. Chronic hepatitis B, chronic hepatitis C, or HIV infection.
3. History of latent or active tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening.
4. Herpes zoster infection within 3 months before randomization
5. Any of the following medications within 6 months of Day 1: cyclophosphamide, leflunomide > 20 mg/day, abatacept.
6. Receipt of a mAb within 5 published half-lives prior to Day 1.
7. Receipt of rituximab or an experimental B-cell depleting mAb within 6 months of Day 1.
8. Receipt of rituximab or an experimental B-cell depleting mAb without return of CD19 or CD20 count to above the lower limit of normal.
9. Receipt of alemtuzumab, bone marrow transplantation, stem cell transplantation, total lymphoid irradiation, or T-cell vaccination therapy -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event | Day 85
  The safety and tolerability of MEDI7734 as measured by the incidence of any adverse events that occur on or after the day of administration of investigational product through the end of follow-up. Laboratory measurements, vital sign measurements, and electrocardiogram (ECG) parameters will also be evaluated as part of safety.

SECONDARY OUTCOMES:
Anti-drug antibodies | Day 85
  Presence of anti-drug antibodies (ADA)
Pharmacokinetics Cmax | Day 85
  Maximum concentration of drug achieved
Pharmacokinetics Tmax | Day 85
  Time at which maximum concentration of drug is achieved
Pharmacokinetic | Day 85
  Half Life
Pharmacokinetic | Day 85
  AUC
Pharmacodynamics | Day 85
  Blood levels of plasmacytoid cells.

OTHER OUTCOMES:
Type I Interferon signature | Day 85
  Neutralization ratio of the type I IFN signature

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Danbury, Connecticut
  - Research Site, DeBary, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. Additional information can be found on astrazenecaclinicaltrials.com.